CLINICAL TRIAL: NCT04145583
Title: A Single-Center, Open-Label, Randomized, Two-Stage, and Two-Way Crossover Study Evaluating Drug-Drug Interaction (DDI) Between HSK3486 Injectable Emulsion and Voriconazole Tablets in Healthy Subjects
Brief Title: A Study Evaluating Drug-Drug Interaction (DDI) Between HSK3486 Injectable Emulsion and Voriconazole Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-107
Record Dates: First submitted 2019-10-25; First posted 2019-10-30 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): 0.4 mg/kg
  Interventions: Drug: HSK3486
- voriconazole , HSK3486 (Experimental): 400 or 200 mg; 0.4 mg/kg
  Interventions: Drug: voriconazole +HSK3486

INTERVENTIONS:
Drug: HSK3486 — Sequence 1: Intravenously infuse 0.4 mg/kg HSK3486 in the morning on an empty stomach. Complete infusion within 1 min.
  Arms: HSK3486
Drug: voriconazole +HSK3486 — Sequence 2: voriconazole：Day 1,400mg，BID；Day 2--Day 6,200mg，BID；200 mg of voriconazole were taken orally in the morning on an empty stomach of Day 7; followed by 1 min intravenous infusion of 0.4 mg/kg HSK3486 30 min later.
  Arms: voriconazole , HSK3486

SUMMARY:
This is a single-center, open-label, randomized, two-stage, two-way crossover study evaluating the effect of voriconazole on the PK, PD, and safety of HSK3486 in healthy subjects.

DETAILED DESCRIPTION:
After the recruited healthy subjects passed the screening of inclusion and exclusion criteria, a seed number was set in the PLAN program of the SAS 9.4 software by the statistician before the formal enrollment, and the subject screening numbers were randomly assigned to the two groups by using a 1:1 block randomization method. The enrolled subjects were assigned a subject number according to the results of randomization and received stage I dosing of HSK3486 injectable emulsion (sequence 1) or HSK3486 injectable emulsion + voriconazole (sequence 2). After a 7-day (sequence 1) or 14-day washout period (sequence 2), the stage II dosing of HSK3486 injectable emulsion + voriconazole (sequence 2) or HSK3486 injectable emulsion (sequence 1) was carried out in a crossover fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females with full capacity for civil conduct, aged ≥18 and ≤45 years old. Both male and female subjects should be enrolled;
2. Male subjects should weigh ≥50 kg, female subjects should weigh ≥45 kg, and the body mass index (BMI) should be ≥19.0 and ≤26.0 kg/m2;
3. Blood pressure should be between 100-140/60-90 mmHg; heart rate should be between 60-99 bpm; body temperature (ear temperature) should be between 35.5-37.1°C; respiration rate should be between 12-20 breaths per minute; SpO2 when inhaling should be ≥95%;
4. Normal results for physical examinations, laboratory tests (blood routine, blood biochemistry, urine routine, and blood coagulation routine), 12-lead electrocardiogram (ECG), chest X-ray, and abdominal B-ultrasound (liver, gallbladder, pancreas, spleen and kidney), or abnormal results without clinical significance as judged by the investigator; no significantly potential difficult airway (modified Mallampati score I-II);
5. No previous history of major organ primary diseases, such as liver, kidneys, digestive tract, blood, metabolic, and cardiovascular diseases; no history of malignant hyperthermia and other genetic conditions; no history of mental/neurological diseases; no history of epilepsy; no contraindications for deep sedation/general anesthesia; no clinically significant history of anesthesia accidents;
6. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with the clinical trial protocol.

Exclusion Criteria:

1. Known allergy to excipients in HSK3486 injectable emulsion (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate, and sodium hydroxide) or voriconazole, or contraindications mentioned in the prescribing information of voriconazole ;
2. In receipt of any one of the following medications or treatments during screening/baseline:

   History of drug abuse or any signs of chronic benzodiazepines use (such as insomnia, anxiety, spasms) within 3 months prior to screening, or a positive urine drug test during baseline; Participated in clinical trials involving any medications or medical devices within 3 months prior to screening, or subjects who have participated in 3 or more drug clinical trials within the past year; In receipt of voriconazole within 4 weeks prior to screening; In receipt of propofol, other sedatives/anesthetics and/or opioid analgesics or compounds containing analgesics within 1 week prior to baseline; In receipt of prescription drugs, Chinese herbal medicines, over-the-counter drugs or food supplements (such as vitamins and calcium supplements) other than contraceptives, paracetamol, oral non-steroidal anti-inflammatory drugs, topical over-the-counter preparations, within 2 weeks prior to baseline; in receipt of strong inhibitors/inducers of CYP enzyme within 7 days prior to baseline, or in receipt of moderate/weak inhibitors/inducers of CYP enzyme within 3 days prior to baseline (see Attachment 4 for the inhibitors and inducers); unless the principal investigator (PI) and the sponsor agree that the medication has no effect on the safety and PK/PD results of the trial.
3. A history or evidence of any one of the following diseases prior to screening/baseline:

   History of cardiovascular diseases such as: Uncontrolled hypertension [SBP ≥170 mmHg and/or DBP ≥105 mmHg without antihypertensive treatment, or SBP >160 mmHg and/or DBP >100 mmHg despite antihypertensive treatment], postural hypotension, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medication, II-III degree atrioventricular block (excluding patients with pacemakers), or QTcF interval ≥450 ms (Fridericia's correction formula); Respiratory insufficiency, history of obstructive pulmonary disease, history of asthma, sleep apnea; history of failed tracheal intubation; history of bronchospasm requiring treatment within 3 months prior to screening; acute respiratory infection, and with obvious symptoms such as fever, wheezing, nasal congestion, or cough within 1 week prior to baseline; History of GI tract diseases: Gastrointestinal obstruction, active GI bleed, potential for reflux and aspiration; Serious infection, trauma, or major surgery within 4 weeks before screening; or acute disease with clinical significance (determined by the investigator) within 2 weeks before screening, including GI diseases or infections (such as respiratory or CNS infections); History of eye diseases: Including glaucoma history and/or family history, history and/or family history of optic nerve diseases, subjects with proliferative diabetic retinopathy, history of intraocular surgery (cataract, retina, glaucoma), history of amblyopia, history of high myopia (≥8.0 D).
4. Laboratory results that meet any of the following during screening/baseline:

   Positive result for either HBsAg, HCV, HIV, or syphilis; Abnormality in any of the following indicators of hepatic and renal functions: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1 x ULN; creatinine > 1 x ULN; total bilirubin TBIL > 1 x ULN;
5. History of alcohol abuse within 3 months prior to screening, abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with40% alcohol or 150 mL wine), or positive result for breath alcohol test (≥20 mg/dl);
6. Smoke more than 5 cigarettes per day and a total of more than 60 cigarettes within 3 months prior to screening;
7. Blood donation or blood loss ≥200 mL within 30 days prior to screening; plasma donation or plasma exchange within 7 days prior to screening;
8. Subjects who consume any beverages or food containing alcohol, grapefruit juice or methylxanthine (such as coffee, tea, coca-cola, chocolate, functional drinks), participate in strenuous physical activities and other factors that may affect drug absorption, distribution, metabolism, and excretion within 2 days prior to enrollment; subjects who are unable to fast for 8 h prior to dose administration;
9. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-05-09 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | From the start of HSK3486 administration to 24 hours after the start of administration on day 1
Area under the concentration-time curve (AUC0-t, AUC0-∞) | From the start of HSK3486 administration to 24 hours after the start of administration on day 1]

SECONDARY OUTCOMES:
Terminal elimination half-life (t1/2) | From the start of HSK3486 administration to 24 hours after the start of administration on day 1

OTHER OUTCOMES:
MOAA/S(modified observer's assessment of alert /sedation) | -5 minutes before administration until 1 hours post administration on day 1
  Observe the change of modified observer's assessment of alert /sedation during the whole trial.
Bispectral index(BIS) | -5 minutes before administration until 1 hours post administration on day 1
  Observe the changes of bispectral index during the whole trial.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Study Director — Medical Ethics Committee of the First Affiliated Hospital of soochow University
Locations (1):
- the First Affilicated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: Undecided